CLINICAL TRIAL: NCT02927782
Title: Flat Bed Rest vs. Immediate Mobilisation After Incidental Durotomy During Lumbar Spinal Surgery: A Prospective Randomised Trial
Brief Title: Mobilisation Algorithm After Incidental Durotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Mazda Farshad, MD MPH, Balgrist University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W569
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-06

CONDITIONS: Cerebrospinal Fluid Leak
Keywords: Cerebrospinal Fluid Leak; Lumbar
MeSH Terms: conditions — Cerebrospinal Fluid Leak | interventions — Early Ambulation; Bed Rest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bed Rest (Active Comparator): 48 hours of strict bed rest after incidental durotomy during lumbar spinal surgery
  Interventions: Procedure: Bed Rest
- Early Mobilization (Experimental): Immediate Mobilization after incidental durotomy during lumbar spinal surgery
  Interventions: Procedure: Early Mobilization

INTERVENTIONS:
Procedure: Early Mobilization — early postoperative mobilisation (walking and sitting). Initial postoperative mobilisation is going to be under supervision of a qualified physiotherapist. The presence of a qualified physiotherapist at first mobilisation is solely for reasons of safety. No specific exercise or regimen is planned.
  Arms: Early Mobilization
Procedure: Bed Rest — 48 hours of strict bed rest followed by postoperative mobilisation under supervision of a qualified physiotherapist. During the bed rest period elevation of the head is tolerated to a maximum of 30°.
  Arms: Bed Rest

SUMMARY:
Patients with persistent symptoms of cerebrospinal-fluid leakage (positional headache, photophobia, nausea and vomiting, clear drainage from the wound, fluctuant subcutaneous wound) after a primary repair should be considered for revision surgery to avoid potentially serious complications including CSF (cerebro spinal fluid) fistula formation. Prolonged bed rest immediatel after reapir of an ID () incidental durotomy) is widely accepted and frequently applied. current literature provides supporting retrospective evidence that prolonged bed rest may not be required after watertight closure of dural tears.

The purpose of this study is to further investigate the impact of prolonged bed rest on the need for early reoperation following primary repair of an ID after lumbar spinal surgery. The primary endpoint of this study is the difference in reoperation rate between the two study groups to further investigate if either one or the other postoperative mobilisation regimen provides a significant benefit in terms of persistent dural leakage.

DETAILED DESCRIPTION:
Patients with persistent symptoms of cerebrospinal-fluid leakage (positional headache, photophobia, nausea and vomiting, clear drainage from the wound, fluctuant subcutaneous wound) after a primary repair should be considered for revision surgery to avoid potentially serious complications including CSF (cerebro spinal fluid) fistula formation.

In a recent retrospective case series of 42 patients Radcliff et al. reported an increase in medical complications including pneumonia and wound infections associated with prolonged bed rest Current literature does not provide prospective nor retrospective evidence on the influence of early mobilization on complications or reoperation rate after ID (incidental durotomy).

Prolonged bed rest is widely accepted and frequently applied after ID. Contrarily, current literature provides supporting retrospective evidence that prolonged bed rest may not be required after watertight closure of dural tears.

The purpose of this study is to further investigate the impact of prolonged bed rest on the need for early reoperation following primary repair of an ID after lumbar spinal surgery. The primary endpoint of this study is the difference in reoperation rate between the two study groups to further investigate if either one or the other postoperative mobilisation regimen provides a significant benefit in terms of persistent dural leakage.

This study is designed as an unblinded, prospective randomised cohort trial. The treatment arms consist of either strict prolonged bed rest for 48 hours or immediate postoperative mobilisation. Patients are going to be randomised into either treatment arm after intraoperative verification of ID. Randomization into either treatment arm is going to be performed in a consecutive alternating manner. The according mobilisation regimen is going to be prescribed by the surgeon performing the index procedure immediately after wound closure as a standard option in the institutions proprietary hospital information system. Symptoms of persisting liquor leakage are going to be assessed by Investigator. Additional confirmation via MRI scan is routinely performed if persistent leakage is suspected and revision surgery is planned. For Patients with symptoms of persisting dural leakage after a 48 hours course of early mobilization a course of 24 hours of bed rest will be administered before revision surgery is scheduled.

Various case series, as well as large pro- and retrospective studies have been published describing incidence, intraoperative management as well as long- and short term outcome of ID. In addition, current literature provides retrospective evidence and small case series considering benefit and adverse events of prolonged bed rest after primarily recognised and repaired ID. To our knowledge this is the first prospective randomised trial to further investigate the impact of immediate mobilisation on the incidence of persistent cerebrospinal leakage.

ELIGIBILITY:
Inclusion Criteria:

All patients over the age of 18 years with an ID sustained during a primary or revision lumbar spinal procedure at our institution are the subject of this prospective, randomised analysis.

Exclusion Criteria:

Patients referred for repair of an externally sustained ID, cases in which durotomy was not primarily recognised and repaired as well as patient who refuse to sign informed consent are going to be excluded from this analysis. Informed consent is going to be obtained one day prior to index procedure.

Further Intervention because of Spondylitis/Spondylodiscitis, Tumor, Trauma. Pregnant patients

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Reoperation rate | 6 weeks
  The primary endpoint of this study is the difference in reoperation rate between the two study groups to further investigate if either one or the other postoperative mobilisation regimen provides a significant benefit in terms of persistent dural leakage.

CONTACTS AND LOCATIONS:
Overall Officials: Mazda Farshad, MD MPH, Principal Investigator — University Hospital Balgrist Zurich
Locations (1):
- University Hospital Balgrist, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No